CLINICAL TRIAL: NCT01018147
Title: 4D Image-guided Adaptive Radiotherapy for Lung Cancer: Patient Image Acquisition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MCC-10395; HM-10395 (Other: VCU IRB); CDR0000657239 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01700 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT Imaging (Experimental): Patients undergo 4-D, 4-dimensional computed tomography, CT imaging prior to radiotherapy sessions and once a week at the end of treatment.
  Interventions: Procedure: 4-dimensional computed tomography

INTERVENTIONS:
Procedure: 4-dimensional computed tomography — Undergo 4-D CT imaging
  Other Names: 4D-CT

SUMMARY:
This clinical trial studies 4-dimensional (4-D) image-guided radiation therapy treatment planning in patients with stage I-IV non-small cell lung cancer. Computed tomography (CT) scans and treatment-planning systems may help in planning radiation therapy for patients with non-small cell lung cancer. This is not a therapy study. Therefore no direct benefit from participating is expected. However, at the discretion of the treating physician, the information gained from the additional imaging will be used to improve treatment accuracy. No patient outcome data are gathered or analyzed by this study. This study is not a:Phase I, II, or III trial, trial with "blinded" treatment arm, gene or a vaccine trial, or a multi-institutional trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Quantify the magnitude and distribution of inter- and intrafraction anatomic variations, including the temporal stability of the tumor/respiration signal correlation.
* Improve the acquisition and reconstruction of 4D CT scan images by advancing the 4D CT scan data collection process and evaluating 4D CT scan image reconstruction using different respiratory inputs.
* Quantify the uncertainty of deformable image-registration algorithms.
* Develop and investigate the efficacy of inter- and intrafraction probabilistic planning-based 4D image-guided adaptive radiotherapy (IGART) strategies for clinical application.
* Determine the expected geometric, dosimetric, and radiobiological improvements from the 4D IGART system.

OUTLINE: Patients undergo insertion of ≥ 1 small radio-opaque marker into (or in the vicinity of) the primary lesion or suspect lymph nodes via bronchoscopy. X-rays are performed to document the position of the markers.

Patients undergo 4D CT scan before each radiotherapy session and once a week after a radiotherapy session. Patients also undergo x-ray imaging before and during radiotherapy, optical and internal marker motion recording before and after radiotherapy, and audiovisual feedback during radiotherapy.

Patients undergo image-guided adapted radiotherapy based on these data.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of non-small cell lung cancer stages I-IV
* Partial pressure oxygen (pO2) > 92%-obtained at the time of or within 3 months prior to initial consultation with the radiation oncologist
* Tumor(s) must be visualized on a CT
* Positron emission tomography (PET) is performed during staging or treatment planning process
* All patients must be informed on the investigational nature of this study and must give informed consent in accordance with institutional guidelines

Exclusion Criteria:

* Pregnant women may not participate; women of reproductive potential must be informed of the need to practice an effective contraceptive method
* Unstable coronary artery disease
* Uncorrectable coagulopathy
* Severe pulmonary hypertension
* Poor tolerance of conscious sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-09; Primary Completion 2012-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
At least 1 mm reduction in overall systematic error corresponding with ≥ 2 mm CTV-PTV margin reduction | Up to 7 years
At least 5 Gy reduction in mean lung dose | up to 7 years
At least 5% reduction in absolute pneumonitis risk (≥ grade 2) | up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F. Williamson, PhD, Principal Investigator — Massey Cancer Center

REFERENCES:
- See also: published article — http://www.pubfacts.com/detail/21626948/A-method-for-robust-segmentation-of-arbitrarily-shaped-radiopaque-structures-in-cone-beam-CT-project
- See also: published article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3354576/
- See also: published article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3259614/
- See also: This article has been featured in: http://biomedfrontiers.org/cancer-2014-2-4/ — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3895914/
- See also: published article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3647023/
- See also: published article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3702591/
- See also: published article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3895914/
- See also: published article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3978354/
- See also: published article — https://ro-journal.biomedcentral.com/articles/10.1186/s13014-015-0435-3